CLINICAL TRIAL: NCT00111436
Title: An Open-Label, Long-Term Extension Study to Assess the Safety of Etanercept in the Treatment of Psoriasis in Adult Subjects
Brief Title: Evaluating the Safety of Etanercept in the Treatment of Psoriasis in Adult Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20030115
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Psoriasis
Keywords: Psoriasis, adults, skin; Phase 3, clinical trial; Amgen, etanercept; Enbrel®, moderate; severe, extension
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular | interventions — Etanercept

ARMS (2):
- 50 mg (Experimental): 50 mg once weekly
  Interventions: Drug: Etanercept
- 100 mg (Experimental): 50 mg twice weekly
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Enbrel 50 mg once weekly or 50 mg twice weekly

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of long-term administration of etanercept in adults with psoriasis who have participated in previous etanercept psoriasis studies. This study will also evaluate the maintenance of the efficacy of etanercept in adults with psoriasis who have participated in previous etanercept psoriasis studies. All subjects enrolled in this study will receive 50 mg once weekly or twice weekly (if qualified after week 12) by subcutaneous injections for at least 48 weeks and up to 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Subjects who were randomized and received at least one dose of investigational product in Study 20021639 or 20021642 (provided that they meet all inclusion/exclusion criteria of this protocol)

Exclusion Criteria:

* Active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit
* Pregnant or breast-feeding females
* Evidence of skin conditions at the time of the screening visit (e.g., eczema) that would interfere with evaluations of the effect of the investigational product on psoriasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2003-04; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events, including infectious episodes | 72 weeks
Changes from baseline in laboratory values | 72 weeks

SECONDARY OUTCOMES:
Improvement in Psoriasis Area and Severity Index (PASI) Score in this study relative to baseline in the original study | 72 weeks
Proportion of subjects who achieve 0 or 1 (clear or almost clear) in the Physician Global Assessment of psoriasis | 72 weeks
Patient Global Assessment of psoriasis | 72 weeks
Percent improvement from baseline in the Dermatology Life Quality Index (DLQI) scores | 72 weeks
Changes from baseline in SF-36 Health Survey scores | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Elewski B, Leonardi C, Gottlieb AB, Strober BE, Simiens MA, Dunn M, Jahreis A. Comparison of clinical and pharmacokinetic profiles of etanercept 25 mg twice weekly and 50 mg once weekly in patients with psoriasis. Br J Dermatol. 2007 Jan;156(1):138-42. doi: 10.1111/j.1365-2133.2006.07585.x. PMID 17199580
- [Result] Leonardi C, Strober B, Gottlieb AB, Elewski BE, Ortonne JP, van de Kerkhof P, Chiou CF, Dunn M, Jahreis A. Long-term safety and efficacy of etanercept in patients with psoriasis: an open-label study. J Drugs Dermatol. 2010 Aug;9(8):928-37. PMID 20684143
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20030115.pdf